CLINICAL TRIAL: NCT01065844
Title: A Phase II Trial of the HIV Protease Inhibitor Nelfinavir in Patients With Recurrent Symptomatic Adenoid Cystic Cancers of the Head and Neck
Brief Title: Nelfinavir in Recurrent Adenoid Cystic Cancer of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: Holden Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, John M. Buatti, Professor & Chair of Radiation Oncology, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200905704
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Results first posted 2016-12-19 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-09

CONDITIONS: Carcinoma, Adenoid Cystic; Head and Neck Neoplasms
Keywords: Nelfinavir
MeSH Terms: conditions — Carcinoma, Adenoid Cystic; Head and Neck Neoplasms | interventions — Nelfinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nelfinavir (Experimental): 1250 mg Nelfinavir twice daily Monday-Sunday
  Interventions: Drug: Nelfinavir

INTERVENTIONS:
Drug: Nelfinavir — 1250 mg Nelfinavir twice daily Monday - Sunday

SUMMARY:
The purpose of this study is to evaluate the FDA-approved drug nelfinavir (NFV) as an oncologic agent for adenoid cystic cancers of the head and neck.

Specifically, subjects will be asked to take 1250 mg twice daily and follow-up with their medical oncologist as clinically indicated while taking this medication.

Subjects would be evaluated for quality of life issues utilizing the EORTC QLQ-C30 2-page questionnaire.

Subjects would also be evaluated clinically by the oncologist to determine if the NFV was having an anti-neoplastic effect.

The study remains unfunded. Therefore, potential subjects must be willing to provide self-travel to study site. This study requires a screening visit, initial study visit, and monthly follow-up. Subjects are not reimbursed for time, travel, or physician costs.

DETAILED DESCRIPTION:
The hypothesis of this study is that nelfinavir, by inhibiting the Akt and MAPK pathways, can inhibit adenoid cystic carcinoid growth. These cancers are heavily dependent on these signalling pathways.

Adenoid cystic carcinomas (ACC) are rare and account for about 1% of all head and neck cancers. They stem from salivary glands and are known for their tendency to spread along nerve sheaths (perineural spread). ACC is known for its prolonged clinical course, multiple recurrence and the delayed onset of distant metastases. The median/mean age at presentation is 47-56. Although 5 year disease free survivals (DFS) are 65-70%, the 15 year DFS drops to 30-40%. If followed long enough, 35% of patients will eventually develop metastatic disease.

The most common treatment of ACC is surgery followed by post-operative radiotherapy. When ACC recurs, management options are often limited both by the morbidity and low efficacy of re-irradiation and repeated surgical resection. Reported response rates to chemotherapy are low and when it occurs, the duration of the response is short lived.

In an effort to explore possible targeted therapies for patients with recurrent ACC, Dr. Gupta's lab examined the activation of 3 signaling proteins (EGFR, Akt, and MAPK) in 9 different paraffinized tissue blocks. Initial indications from in vitro studies demonstrates NFV is tumoricidal at clinically achievable concentrations. To explore the clinical benefit of this FDA-approved medication, we seek to implement its off label use in patients who have failed all other therapies and have no other therapeutic options left.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of adenoid cystic carcinoma.
* Cancer should be staged recurrent or end-stage with/without metastases who have failed all other therapy.
* Age ≥ 18 years
* ECOG performance status 0-2 (Karnofsky ≥ 50%, see Appendix A).
* Patients must have normal organ and marrow function as defined below:

  * leukocytes ≥ 3,000/mm3
  * absolute neutrophil count ≥ 1,500/mm3
  * platelets ≥ 100,000/mm3
  * total bilirubin < 1.5 mg/dl OR a stable or a decreasing bilirubin in patients who have undergone placement of an intrabiliary stent
  * AST(SGOT) ≤ 2.5 X institutional upper limit of normal
  * ALT(SGPT) ≤ 2.5 X institutional upper limit of normal
  * creatinine < 1.5 X institutional upper limit of normal OR creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
* No known HIV infection. Since NFV is used in HIV patients, we do not want to interfere with the therapy the patient may already be on.
* Not pregnant. The effects of NFV on the developing human fetus have been studied in HIV positive women (21). We do not, however, know the risks along with radiation. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to NFV.
* Uncontrolled diabetes.
* Hemophilia A & B as increased bleeding during protease inhibitor therapy has been reported (22).
* Patients may not be receiving any other investigational agents. concomitant medications counterindicated for use with nelfinavir
* Pregnant or lactating women: The effects of NFV on the developing human fetus have been studied in HIV positive women (21). In addition, the chemotherapy will be deleterious to the fetus.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with NFV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M. Buatti, M.D., Principal Investigator — University of Iowa
Locations (1):
- The Holden Comprehensive Cancer Center, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta AK, Wilke WW, Taylor EN, Bodeker KL, Hoffman HT, Milhem MM, Buatti JM, Robinson RA. Signaling pathways in adenoid cystic cancers: implications for treatment. Cancer Biol Ther. 2009 Oct;8(20):1947-51. doi: 10.4161/cbt.8.20.9596. Epub 2009 Oct 22. PMID 19729990
- [Result] Hoover AC, Milhem MM, Anderson CM, Sun W, Smith BJ, Hoffman HT, Buatti JM. Efficacy of nelfinavir as monotherapy in refractory adenoid cystic carcinoma: Results of a phase II clinical trial. Head Neck. 2015 May;37(5):722-6. doi: 10.1002/hed.23664. Epub 2014 Jun 18. PMID 24596143

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nelfinavir
Started | 15
Completed | 10
Not Completed | 5
Not completed — Adverse Event | 5

BASELINE CHARACTERISTICS:
Arm/Group | Nelfinavir
Number analyzed (Participants) | 15
Age, Customized [Count of Participants; unit: Participants] — Age, in years, of study participants at consent
  Participants
    <=18 years | 0
    Between 18 and 65 years | 12
    >=65 years | 3
Sex/Gender, Customized [Count of Participants; unit: Participants] — Self-reported gender at time of study enrollment
  Participants
    Female | 9
    Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Tumor Progression
Description: Tumor progression as defined by RECIST version v1.1 criteria with ordinal measurements of complete response (CR), partial response (PR), stable disease (SD), and progressive disease (PD).
Time Frame: Every 1 to 3 months
Population: Those with adverse events necessitating interruption of intervention and removal from study were not assessed for outcome measures
Measure: Count of Participants; unit: Participants
Arm/Group | Nelfinavir
Number analyzed (Participants) | 11
Participants
  Complete reponse (CR) | 0
  Partial response (PR) | 0
  Stable disease (SD) | 7
  Progressive disease (PD) | 4

ADVERSE EVENTS:
Time Frame: Adverse event data collected from day 1 of nelfinavir therapy through 30 days after final nelfinavir dose.
Arm/Group | Nelfinavir
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 5/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nelfinavir (N=15)
platelet count decreased (Blood and lymphatic system disorders) | 1 (1) — grade 3
dizziness, grade 3 (Nervous system disorders) | 1 (1) — A disorder characterized by a disturbing sensation of lightheadedness, unsteadiness, giddiness, spinning or rocking. Grade: Severe - limiting activities of daily life
hyponatremia, grade 4 (Metabolism and nutrition disorders) | 1 (1) — A disorder characterized by laboratory test results that indicate a low concentration of sodium in the blood.
Investigations - Other, liver enzymes increased, grade 3 (Investigations) | 2 (2) — Marked elevations across liver function tests considered severe (grade 3)

LIMITATIONS AND CAVEATS:
Favorable selection criteria were used in study design. RECIST assessed at a median interval of 12 weeks - this difference in methods may have artificially prolonged the progression free survival observed in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes